CLINICAL TRIAL: NCT00635011
Title: Pre- and Postoperative Cognitive Behavior Therapy for Patients Accepted for Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Fonna (Other)
Collaborators: Helse Vest (Other)
Responsible Party: Principal Investigator, Haldis Økland Lier, PhD, medical doctor, Helse Fonna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16280
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Obesity, Morbid
Keywords: comorbidity; Quality of Life; Body Weight Changes
MeSH Terms: conditions — Obesity, Morbid; Body Weight Changes | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: psychotherapy — Cognitive Behavioral therapy

SUMMARY:
The purpose of this study is to investigate the relationship between the potential predictive psychological variables and success after bariatric surgery. The investigators will also investigate the purpose of a pre- and postoperative psychological intervention.

DETAILED DESCRIPTION:
Bariatric surgery is the treatment of choice for morbid obesity, but it does not lead to equal results in every patients. Research about personality factors involved in successful outcome after bariatric surgery has led to contrasting results. The existing literature about potential predictors of success after bariatric surgery is far from conclusive. The investigators want to evaluate preoperatively by standardized diagnostic interviews (MINI, SCID-II) and rating scales and questionnaires to assess co-morbid psychopathology. The same evaluation will be done after 1,2 and 5 years. The investigators will look for a relationship between psychological variables and success after bariatric surgery, including amount of weight loss, psychiatric comorbidity, quality of life and employment. The investigators will also investigate the purpose of an pre- and postoperative psychological intervention. Patients on a waiting list for bariatric surgery are randomised to an intervention- and a control group. The intervention is based on cognitive behavior therapy and mindfulness, 6 weeks preoperative and two weeks postoperative programme. Outcome measures are amount of weight loss, psychiatric comorbidity, quality of life and employment.

ELIGIBILITY:
Inclusion Criteria:

* Patients on a waiting list for bariatric surgery at Haugesund hospital

Exclusion Criteria:

* Patients with psychosis and suicidality
* Suicidal attempts the last two years
* Or suicidal thoughts or plans.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
psychiatric comorbidity | five years

SECONDARY OUTCOMES:
weight loss | five years

CONTACTS AND LOCATIONS:
Overall Officials: Haldis Oe Lier, MD, Principal Investigator — Haugesund Hospital, Helse Fonna HF
Locations (1):
- Haugesund Hospital, Helse Fonna HF, Haugesund, Rogaland, Norway

REFERENCES:
- [Result] H.Ø.Lier, E. Biringer, H. Eriksen, T. Tangen. Subjective health complaints in a sample with morbid obesity and the complaints' relation with work ability. Poster presentation, 17 th European congress of psychiatry, January 24-28, 2009- Lisbon, Portugal
- [Result] Lier HO, Biringer E, Stubhaug B, Eriksen HR, Tangen T. Psychiatric disorders and participation in pre- and postoperative counselling groups in bariatric surgery patients. Obes Surg. 2011 Jun;21(6):730-7. doi: 10.1007/s11695-010-0146-7. PMID 20396993
- [Result] Lier H, Biringer E, Stubhaug B, Eriksen HR, Tangen T. Patient outcome expectancy from bariatric surgery. European Psychiatry 25 (supplement 1), 2010 819. 18 th European Congress of Psychiatry. February 27, March 2, 2010-Munich, Germany
- [Derived] Lier HO, Biringer E, Hove O, Stubhaug B, Tangen T. Quality of life among patients undergoing bariatric surgery: associations with mental health- A 1 year follow-up study of bariatric surgery patients. Health Qual Life Outcomes. 2011 Sep 26;9:79. doi: 10.1186/1477-7525-9-79. PMID 21943381